CLINICAL TRIAL: NCT01582919
Title: STUDY OF IMAGING MARKERS IN THE VERY EARLY STAGES OF DEMENTIA AMONG RETIRED RURAL FARM IN THE GIRONDE AND PARTICIPATING IN THE AMI COHORT EPIDEMIOLOGY: A LONGITUDINAL STUDY.
Brief Title: Neuroimaging Markers of Alzheimer Disease: a Longitudinal Population Study
Acronym: AMIMAGE 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2011/15
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Dementia; Alzheimer Disease
Keywords: dementia; Alzheimer's Disease; diagnostic; biomarkers; neuroimaging; PET; MRI; mild cognitive impairment
MeSH Terms: conditions — Dementia; Alzheimer Disease; Disease; Cognitive Dysfunction | interventions — Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participant from AMI cohort (Experimental)
  Interventions: Other: Neuroimaging
- Participant from 3Ccohort (Active Comparator)
  Interventions: Other: Neuroimaging

INTERVENTIONS:
Other: Neuroimaging

SUMMARY:
It is now acknowledged that Alzheimer's disease is characterized by a long period of pathophysiological change. Developing new strategies to achieve diagnoses as early as possible has become a major goal for therapies aimed at slowing the progression of this disease. While diagnoses currently rely principally on clinical neuropsychology, the typical diagnostic criteria of NINCDS-ADRDA are inapplicable in the early stage of the disease. The goal of our project is to identify very early imaging markers for Alzheimer's disease among patients with no report of cognitive difficulties. In order to achieve this goal, we propose a longitudinal study in an elderly population cohort.

DETAILED DESCRIPTION:
The AMImage2 project that follows AMImage1 and MRI-3C consists of an imaging study in association with longitudinal epidemiologic cohorts (AMI and 3C). The first objective is to investigate the association between the evolution of imaging markers and the evolution of cognitive performance in normal and pathological aging. This objective will be conducted among subjects having already participated in AMImage1, thereby permitting the longitudinal study of MRI data. An MRI exam will also be proposed to 100 subjects (members of the AMI and 3C cohorts) in order to provide a third wave of MRI (for a longer-term MRI follow-up) or a second one for the participants who only had one MRI exam in the AMImage project. Our second objective is cross-sectional and will study the imaging parameters of subjects presenting signs of cognitive decline over the previous 4 years (through the follow-up conducted in the AMI cohort). Finally, an additional objective will consist in a comparison between two populations very contrasted in terms of cognitive reserve: AMI (very low education level in rural area) and 3C (higher level of education in urban area).

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years old
* Be retired from agricultural profession
* live in rural area in Gironde (France)

Exclusion Criteria:

* Lefthanded
* having a dementia (MMSE < 13)
* Having a vascular cerebral accident
* Parkinson disease
* RMI exclusion criteria
* [18F]-FDG PET SCAN exclusion criteria
* Poor health condition does not allowing transport to neuroimaging service

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 304 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Measures of volume and diffusion parameters in the gray matter (hippocampus and cingular posterior cortex) | Inclusion (Day 0)

SECONDARY OUTCOMES:
Performance on neuropsychological and daily life cognitive tests | Everyday up to Day 7 after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Michèle ALLARD, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Groupe Hospitalier Pellegrin - C.H.U. de Bordeaux, Bordeaux, France